CLINICAL TRIAL: NCT05067374
Title: Screening for the Hepatitis C Virus by TROD Paired With Mammography and Management of Chronic Hepatitis C in Women Aged 50 to 74 in the Agglomeration of Montpellier
Brief Title: Hepatitis C Screening Paired With Mammography
Acronym: Mammo'C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0005-UF7919
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis C; Breast Cancer
Keywords: Rapid orientation diagnostic test; Hepatitis C; Breast cancer; Mammography; Blood sample; Paired screening
MeSH Terms: conditions — Hepatitis C; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France, a breast cancer screening is organized since 2004 for women aged 50-74. On the other hand, even though the seroprevalence of hepatitis C in the general French population is less than 1%, it is estimated that more than 75,000 people live with the virus without knowing it. To answer the WHO objective of eliminating hepatitis C by 2030 and in France by 2025, the investigators need to organize targeted screening. Women aged more than 50 years old, by their possible antecedents in life, are an exposed population. The investigators propose to pair the already organized breast cancer screening with a hepatitis-screening test by rapid diagnostic orientation test (TROD) and evaluate the adherence of women in this paired screening. For women with positive TROD, a specialized care will be organized.

DETAILED DESCRIPTION:
Context :

Organized breast cancer screening has been introduced in France since 2004. It concerns women aged 50 to 74 years old with average risk (no symptoms and no risk factors). This systematic screening reaches approximately 70% of the includable women. At the same time, it is estimated that 10 to 15% of women aged 50 to 74 undergo screening as part of an individual detection process.

The seroprevalence of hepatitis C in the general French population is less than 1%, but it is estimated that around 75,000 people living with the virus are unaware of their seropositivity. Among them, the risk of a late diagnosis is the risk of cirrhosis or hepatocellular carcinoma. Screening for hepatitis C is also justified now that the new treatments is universally accessible with a remarkable efficacy (>95%). These pan-genotypic treatments are of short duration and have very few adverse effects.

The WHO has set a goal of eliminating hepatitis by 2030 and France has gone a step further and proposed an elimination date of 2025. These objectives are not achievable without improved screening, the cornerstone of access to treatment. The objective is therefore to propose targeted screening in certain sub-population to organize micro elimination phenomena. Women over 50 years of age constitute a sub population at risk.

Objectives :

The objective of the study is to evaluate the adherence rate of women aged 50 to 74 years to hepatitis C screening by TROD paired with systematic breast cancer screening.

The secondary objectives of the study are, among women aged 50-74 presenting for breast cancer screening in the city of Montpellier, to estimate:

* The prevalence of viral hepatitis C
* The prevalence of chronic viral hepatitis C
* The retrospective care cascade of hepatitis C in women screened positive for chronic hepatitis C
* Access to hepatitis C care among positive for chronic hepatitis C

Methodology:

Type of study: Prospective screening procedure evaluation study.

Primary endpoint:

- The number of women who agreed to undergo the HCV test among those who were offered the test will be calculated = adherence to the proposed screening.

Secondary endpoints:

* Number of hepatitis C positive TRODs compared to the number of TRODs performed
* Number of HCV RNA positives among the number of hepatitis C positive TRODs.
* Retrospective chronic viral hepatitis C care cascade for participants with a positive TROD
* Access to care and prospective cascade of care

Statistical analysis:

The main analyses will be descriptive. The main characteristics of the participants will be described by the mean/standard deviation or median/interquartile range when the variable is quantitative and by a proportion with confidence interval when the variable is qualitative.

The judgment criteria will be described by percentages with their 95% confidence intervals. The fibrosis score will be presented in classes.

ELIGIBILITY:
Inclusion Criteria:

* - Women aged 50-74 inclusive
* Doing a breast cancer screening
* Able to understand and complete a questionnaire on their own or with the help of a third party
* Able to understand the study and follow the protocol
* Having signed the consent form
* With social security plan

Exclusion Criteria:

* - Cannot sign the consent or follow the protocol
* Under French legal protection measure (sauvegarde de justice, tutelle or curatelle)

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women participating in the organized systematic breast cancer screening
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-03-23 (Estimated); Study Completion 2025-03-23 (Estimated)

PRIMARY OUTCOMES:
Adherence to the hepatitis C screening | At inclusion
  Description: Number of women who have agreed to do the hepatitis C screening by rapid orientation diagnostic test (TROD) among the woman to whom it was offered.

SECONDARY OUTCOMES:
Percentage of positive hepatitis C TROD | At inclusion
  Number of positive TROD among the number of TROD done
Percentage of positive hepatitis C RNA | at 1 year after inclusion day
  Number of positive HCV RNA blood samples among the positive TROD for hepatitis C
Retrospective care cascade : percentage of women with knowledge of their positive serological status | At inclusion day
  Number of women with knowledge of their HCV serological status among women with a TROD
Retrospective care cascade : percentage of women with a HCV viral load done | At inclusion day
  Number of women with a HCV viral load done in the past among the women with knowledge of their positive serological status.
Retrospective care cascade : percentage of treated women | At inclusion day
  Number of women who had already been treated for hepatitis C in the past among women with a positive viral HCV charge.
Retrospective care cascade : percentage of women cured | at 1 year after inclusion day
  Number of women who had already been cured of HCV in the past among the women treated.
Care access and prospective care cascade : percentage of women with a blood test done | At inclusion day
  Number of women with a blood test done among the number of prescriptions given when the TROD is positive
Care access and prospective care cascade : percentage of women with positive HCV RNA | at 1 year after inclusion day
  Number of women with a positive HCV RNA blood test among women with a prescribed blood test
Care access and prospective care cascade : percentage of women who consulted with the hepatologist | At inclusion day
  Number of women who had a consultation with the hepatologist among women with a positive TROD
Care access and prospective care cascade : percentage of women who initiated the treatment | At inclusion day
  Number of women who initiated their treatment among women with a positive HCV RNA in women who had a consultation with the hepatologist
Care access and prospective care cascade : Fibrosis score | At inclusion day
  Fibrosis score of women who had the prescribed blood test done
Care access and prospective care cascade : percentage of cured women | 12 weeks after the end of treatment
  Number of women cured for HCV 12 weeks after the end of treatment among women who initiated the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hélène DONNADIEU RIGOLE, Pr, Principal Investigator — Biochemistry department
Locations (4):
- France (4):
  - Beausoleil private clinic, Montpellier, Occitanie
  - Lapeyronie radiology ward (Montpellier University hospital), Montpellier, Occitanie
  - Le Millénaire private clinic, Montpellier, Occitanie
  - Victor Hugo Center, Montpellier, Occitanie